CLINICAL TRIAL: NCT05568290
Title: Evaluation of Interleukin-38 Levels in Individuals With Healthy and Periodontal Disease
Brief Title: Interleukin-38 Levels in Individuals With Periodontitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Other Study IDs: IstanbulSBU
Record Dates: First submitted 2022-09-10; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-09

CONDITIONS: Periodontitis; Gingivitis; Healthy
Keywords: periodontal disease; IL-38
MeSH Terms: conditions — Periodontitis; Gingivitis; Periodontal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Periodontitis: Individuals with Periodontitis
  Interventions: Other: Saliva; Other: gingival crevicular fluid
- Gingivitis: Individuals with Gingival Inflammation
  Interventions: Other: Saliva; Other: gingival crevicular fluid
- Healthy: Individuals with Periodontally Healthy
  Interventions: Other: Saliva; Other: gingival crevicular fluid

INTERVENTIONS:
Other: Saliva — individuals' saliva samples will be collected and transferred to eppendorf tubes.
  Until biochemical analysis is carried out will be stored in -80ºC.
  Other Names: sampling
Other: gingival crevicular fluid — GCF samples of individuals will be collected by paper strips and transferred to eppendorf tubes.Until biochemical analysis is carried out will be stored in -80ºC.
  Other Names: sampling

SUMMARY:
Interleukin (IL)-38 is the newest member of the IL-1 family. It can bind to receptors through various pathways and regulate the formation and function of inflammatory cytokines. Periodontitis is a chronic inflammatory disease that can start with localized inflammatory reactions created by the supporting tissues surrounding the teeth against microorganisms and then result in loss of teeth. The aim of this study is to compare the IL-38, IL-1β and IL-10 levels of healthy and periodontitis individuals.

DETAILED DESCRIPTION:
Periodontitis is a destructive chronic inflammatory disease that can start with localized inflammatory reactions created by the supporting tissues surrounding the teeth against microorganisms and then result in loss of teeth. More than any other cytokine family, the interleukin (IL)-1 family (IL-1α, IL-1β, IL-18, IL-33, IL-36α, IL-36β, IL-36γ, IL-1Ra, IL-36Ra, IL-37, IL-38) includes key signaling molecules that trigger and perpetuate periodontal inflammation.

Interleukine -1β ( IL-1β ) levels are associated with periodontal destruction in the pathogenesis of periodontal disease. Interleukine-10 (IL-10) has been reported to decrease periodontal disease progression rate.

Gingival crevicular fluid shows the cellular response in the periodontium. The most important host-related ingredients are inflammatory markers, including cytokines, enzymes, and interleukins. Saliva analysis is used in the diagnosis of systemic conditions as well as in the diagnosis of oral pathologies.

In recent studies, IL-38 expression has been reported to be abnormal (abnormal) in chronic inflammatory diseases, especially in rheumatoid diseases such as systemic lupus erythematosus, rheumatoid arthritis, psoriasis, and inflammatory bowel disease. Therefore, this relationship of this inflammatory cytokine with chronic inflammatory diseases draws attention to the regulatory effect of IL-38 in these diseases. The aim of this study is to compare the IL-38, IL-1β and IL-10 levels of healthy and periodontitis individuals.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy individuals who does not have a disease under treatment,
* individuals without regular systemic medication

Exclusion Criteria:

* smoking
* receiving periodontal treatment in the last 6 months
* pregnancy
* lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals will be divided into three different groups, about 20-25 people in each group.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2022-11-10 (Estimated); Study Completion 2022-12-10 (Estimated)

PRIMARY OUTCOMES:
IL-38 levels | initial examination, baseline
  saliva and DOS levels
IL-1β levels | initial examination, baseline
  saliva and DOS levels
IL-10 levels | initial examination, baseline
  saliva and DOS levels

SECONDARY OUTCOMES:
Plaque Index | initial examination, baseline
  Silness-Löe
Probing Depth | initial examination, baseline
  millimeter
Bleeding on Probe | initial examination, baseline
  Ainamo&Bay

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Toraman, Dr, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Saglik Bilimleri Universitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No